CLINICAL TRIAL: NCT00629954
Title: Abuja Heart Study (AHS) is a Multi-site Prospective Epidemiological Investigation of Cardiovascular Disease (CVD) .
Brief Title: Abuja Heart Study: Prospective Epidemiological Investigation of Cardiovascular Diseases
Acronym: AHS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Healthsystem Plus (Other)
Collaborators: Federal Ministry of Health, Nigeria (Other Government); Akaza Research (Industry); Byrne Healthcare (Industry); Baim Institute for Clinical Research (Other)
Responsible Party: Principal Investigator, uchenna onyeachom, Study Director/ Principal Investigator, Healthsystem Plus
Other Study IDs: HIFA-001
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2012-08

CONDITIONS: Cardiovascular Diseases; High Blood Pressure
Keywords: ABUJA HEART STUDY NIGERIA; CARDIOVASCULAR DISEASES
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I

SUMMARY:
This is a multi-site prospective epidemiological investigation of cardiovascular disease (CVD) among Abuja residents from the rural and metropolitan area.

DETAILED DESCRIPTION:
Sub-Saharan Africa continues to fight the battle of infectious diseases such as HIV/AIDS, Tuberculosis and Malaria. But given all the international efforts geared to curing and containing these diseases, and with progress made in various countries, Sub-Saharan Africa is now heading into another type of epidemic, cardiovascular disease (CVD). Predicted statistics have shown that cardiovascular diseases will become the leading cause of death in developing countries within the next 10 to 15 years, however relatively few population-based studies have examined CVD in Africa .

Although control of communicable ,childhood ,and maternal diseases has benefited from an international efforts on clinical care, policy and implementation,such large scale effort are lacking for CVD and have left both policymakers and individuals with decisions on health issues without adequate information.

Prior to the commencement of the study,series of community meetings and focus groups discussions will be held to identify ways to enhance participation. An extensive examination will include a series of questionnaires dealing with lifestyle habits, medical history, social and cultural factors, physical assessments which include height, weight,central blood pressure assessment of arterial stiffness and autonomic function and laboratory measurements for cholesterol, other lipids, glucose ,c-reactive protein among others.

ELIGIBILITY:
Inclusion Criteria:

* Some history of cardiovascular disease,PLWHA
* Patients have to agree to participate by signing a consent
* 18 years and older

Exclusion Criteria:

* Stroke

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Abuja residents from the rural and metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
determine the roles of sociocultural factors, such as poverty,gender, literacy, stress in the development of CVD and associated risk factors | 5

SECONDARY OUTCOMES:
familial or hereditary factors | 10

CONTACTS AND LOCATIONS:
Overall Officials: Uchenna N Onyeachom, Principal Investigator — Healthsystem Plus; Ngozi A Njepuome, Principal Investigator — Abuja Heart Study; Chimele Abengowe, Study Chair — National Hospital, Abuja
Locations (5):
- Nigeria (5):
  - National Hospital Abuja, Abuja, Federal Capital Territory
  - State House Medical Center, Abuja, Federal Capital Territory
  - Bwari General Hospital, Bwari, Federal Capital Territory
  - Nigerian Defense Medical Center, Abuja
  - Gwagwalada Specialist Hospital, Federal Capital Territory